CLINICAL TRIAL: NCT07116525
Title: Clinical Evaluation of Arrhythmia Mapping With a Paddle-shaped, High-density, Multi-electrode Mapping Catheter
Brief Title: A Study Assessing Arrhythmia Mapping With a Multi-Electrode Mapping Catheter
Acronym: FEATHER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BWI202307; BWI202307 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Scar-related Atrial Tachycardia; Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Ventricular Procedures; Ventricular Tachycardia; Ischemic Ventricular Tachycardia; Non-ischemic Ventricular Tachycardia; Cardiomyopathy; Idiopathic Ventricular Tachycardia; Premature Ventricular Contraction
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular; Cardiomyopathies; Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Arrhythmia Mapping by a Paddle-shaped, High-density, Multi-electrode Mapping Catheter (Experimental): Participants scheduled to have a clinically indicated catheter mapping and ablation procedure for management of a cardiac arrhythmias will undergo catheter mapping and ablation procedure using paddle-shaped, high-density, multi-electrode mapping catheter.
  Interventions: Device: Paddle-Shaped, High-Density, Multi-Electrode Mapping Catheter

INTERVENTIONS:
Device: Paddle-Shaped, High-Density, Multi-Electrode Mapping Catheter — High-density, multi-electrode mapping catheter will be used for the procedure.

SUMMARY:
The purpose of this study is to assess the safety and feasibility of the investigational catheter for mapping the atrial and ventricular regions of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with and candidate for clinically indicated catheter mapping and ablation procedure for the management of ventricular tachycardia, premature ventricular complex, atrial tachycardia or atrial fibrillation (participant having undergone a previous ablation procedure may be included)
* At least one episode of the targeted arrhythmia (ventricular tachycardia, premature ventricular complex, atrial tachycardia or atrial fibrillation) must have been documented by electrocardiogram (ECG), Holter, loop recorder, telemetry, implanted device, or transtelephonic monitoring within 12 months prior to enrollment
* Age 18 years or older
* Signed Patient Informed Consent Form (ICF)
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* Study arrhythmia secondary to reversible cause, or secondary to electrolyte imbalance, thyroid disease, or non cardiac cause
* Patients requiring left atrial procedures: left atrial size greater than (>) 55 millimeter (mm)
* Left ventricular ejection fraction(LVEF) less than or equal to (<=) 25 percentage (%) for participants with ventricular arrhythmia
* LVEF <= 40% for participants with atrial arrhythmia
* Documented intracardiac thrombus as detected on imaging within 24 hours prior to insertion of the investigational catheter
* Contraindication to anticoagulation (that is, heparin, warfarin, dabigatran)
* History of blood clotting or bleeding abnormalities (example hypercoagulable state)
* Myocardial infarction within the past 2 months (60 days)
* Documented thromboembolic event (including transient ischemic attack [TIA]) within the past 12 months (365 days)
* Uncontrolled heart failure or New York heart association (NYHA) function class IV
* Implanted with a pacemaker or intracardiac cardiac defibrillator or appendage closure device within the past 6 weeks (42 days)
* Patients with known untreatable allergy to contrast media
* Active illness or active systemic infection or sepsis
* Diagnosed atrial or ventricular myxoma, interatrial baffle or patch, tumor or other abnormality that precludes catheter introduction or manipulation
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Participants that have ever undergone a percutaneous or surgical valvular cardiac procedure (that is, ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
* Participants that currently have Impella or equivalent devices on the procedure date or up to 7 days prior
* Any cardiac surgery within the past 60 days (2 months) (includes percutaneous coronary intervention [PCI])
* Atrial septal closure within the past 6 weeks (42 days)
* Presence of a condition that precludes vascular access
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of childbearing age and plan on becoming pregnant during the course of the clinical investigation
* Categorized as vulnerable population and requires special treatment with respect to safeguards of well-being
* Concurrent enrollment in an investigational study evaluating another device or drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) Within 7 Days of Index Procedure Related to the Investigational Catheter When Used for Endocardial Mapping | Up to 7 days post index procedure
  A SAE is any AE that led to any of the following: (1) Death; (2) Serious deterioration in the health of a participant that resulted in any of the following: Life-threatening illness or injury; Permanent impairment of a body structure or a body function; In-patient hospitalization or prolongation of patient hospitalization; Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to body structure or a body function; Chronic disease. (3) Fetal distress, fetal death or a congenital physical or mental impairment or birth defect.
Incidence of Completion of All Pre-Ablation Endocardial Mapping Requirements and Any Clinically Indicated Endocardial Mapping | Up to 7 days post index procedure
  Incidences of all pre-ablation endocardial mapping requirements and any clinically indicated endocardial mapping with the investigational catheter, without resort to non-investigational mapping catheter due to an inadequacy or inability of the investigational catheter to perform the required arrhythmia mapping will be reported.

SECONDARY OUTCOMES:
Investigator Assessment of Deployment; Visualization; Maneuverability and Signal Quality | Up to 7 days post index procedure
  Physician feedback on the catheter deployment, visualization, maneuverability, and signal quality acquired with the investigational catheter for mapping of the atria and ventricles, inclusive of endocardial and epicardial spaces, using a physician-completed survey, using a Likert scale of 1 to 7 (1=poor and 7=excellent) will be summarized.
Incidence of SAEs Related to the Investigational Catheter When Used for Epicardial Mapping as per Physician's Discretion | Up to 7 days post index procedure
  A SAE is any AE that led to any of the following: (1) Death; (2) Serious deterioration in the health of a participant that resulted in any of the following: Life-threatening illness or injury; Permanent impairment of a body structure or a body function; In-patient hospitalization or prolongation of patient hospitalization; Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to body structure or a body function; Chronic disease. (3) Fetal distress, fetal death or a congenital physical or mental impairment or birth defect.
Incidence of all Other SAEs Not Related to the Investigational Catheter | Up to 7 days post index procedure
  Incidence with all other SAEs not related to the investigational catheter will be reported.
Incidence of Non-serious Adverse Events (AEs) Related to the Investigational Catheter | Up to 7 days post index procedure
  Incidence with non-serious AEs related to the investigational catheter will be reported.
Incidence of Completion of all Pre-ablation Epicardial Mapping Requirements and Any Clinically Indicated Epicardial Mapping With the Investigational Catheter as Per Physician's Discretion | Up to 7 days post index procedure
  Incidence of completion with all pre-ablation epicardial mapping requirements and any clinically indicated epicardial mapping with the investigational catheter as per physician's discretion, without resort to non-investigational mapping catheter due to an inadequacy or inability of the investigational catheter to perform the required arrhythmia mapping will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (6):
- Belgium (2):
  - AZ Sint-Jan, Bruges
  - Jessa Ziekenhuis, Hasselt
- France (3):
  - Hopital les Franciscaines of Nimes, Nîmes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Chu Rennes Hopital Pontchaillou, Rennes
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency